CLINICAL TRIAL: NCT06662305
Title: Vaping Cessation Among Youth: Evaluating the Kick-Nic! App
Brief Title: Kick-Nic! Youth Quit Vaping App
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000035028; 1R01CA285216-01A1 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Nicotine Vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into an ACTIVE group or CONTROL group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIVE (Experimental): Participants in the active group will be given access to the Kick-Nic! app to use for vaping cessation.
  Interventions: Behavioral: Kick-Nic! mobile phone application
- CONTROL (Active Comparator): Participants in the control group will be referred to the NCI Quit Vaping website.
  Interventions: Behavioral: NCI Quit Vaping website

INTERVENTIONS:
Behavioral: Kick-Nic! mobile phone application — The Kick-Nic! app has seven modules that cover core CBT strategies using skills, graphic illustrations, and interactive components to help adolescents quit using e-cigarettes.
  Arms: ACTIVE
Behavioral: NCI Quit Vaping website — The NCI webpage provides quitting tobacco resources for youth, including for e-cigarettes. The information provided is similar to the CBT skills modeled by the Kick-Nic! app.
  Arms: CONTROL

SUMMARY:
High school students who want to quit vaping will be randomized to receive the Kick-Nic! app or a control NCI website to determine the efficacy of the app for vaping cessation. Participants will be screened for eligibility, then go through an 8 week treatment period where they will be given access to use the Kick-Nic! app or referred to the NCI Quit Vaping website. This will be followed by 1, 2, 3, and 6 month follow up visits. Qualitative interviews with participants and school staff will also be conducted to obtain feedback on the app and best ways to implement/disseminate the app.

Abstinence rates will be assessed biweekly during treatment including at end of treatment (EOT), and then at 1, 2, 3 and 6 month follow ups (FU). Biochemical verification (salivary cotinine < 30 ng.ml) of self-reports of abstinence will be conducted at EOT and 6-month FU.

DETAILED DESCRIPTION:
Youth will be randomized to receive the Kick-Nic!© app (ACTIVE group) or a CONTROL assessment condition who will be given referrals to the NCI Quit Vaping webpage.

Description of NCI Quit Vaping webpage: The NCI webpage provides quitting tobacco resources for youth, including for e-cigarettes. Importantly, the information provided is similar to the CBT (Cognitive Behavioral Therapy) skills modeled by the Kick-Nic! © app. The Quit Vaping section provides education/modules on how to quit vaping including 1) "build my quit plan", 2) "get a vaping reality check", 3) "how to quit vaping", 4) "your first day without vaping", 5) "deal with vape cravings", 6) "understand your vape triggers", 7) "vaping addiction and nicotine withdrawal", 8) "anxiety, stress and vaping", and 9) "depression and vaping". Adolescents have the option of speaking to an NCI LiveHelp specialist, and access to a Quitline number (800-QUIT-NOW) which can provide further access to counselors.

ACTIVE group participants will be introduced to the app. They will receive instructions on logging in, navigation and will receive a FAQ sheet (via text or email) that will detail this information. They will receive standard advice to avoid use of other tobacco products, cannabis, or e-cigarettes without nicotine. Participants will be asked to use the app over an 8-week period, complete one module each week, and practice the skills that they learned between modules. They will be told that the app will help them set a quit day and that they should complete the first two modules which would teach them how to prepare for quitting before their quit day.

Engagement will be encouraged using text/motivational messages and weekly personal check-ins. Additionally, participants will also receive weekly personal check-ins during the 8-week treatment period which will be conducted by research staff and will use voice or video calls (preferably) or text (depending on the participant's preference) and a standardized script for various scenarios. Staff will check in on whether participants completed the modules. If not, they will provide support to address any barriers to completing the modules, motivational messages to encourage module completion and to practice skills they will learn. If participants have completed the module that was due to be completed that week, they will receive motivational messages to encourage them to practice the skills they learned. The check-ins will not provide any further quit advice (to avoid interfering with the content of the app).

Assessments will be obtained at baseline (week 0; treatment initiation), every two weeks (weeks 2, 4, 6, 8) during the treatment period, and then at 1, 2, 3 and then 6 months follow up timepoints by research assistants who will be blind to the randomization condition.

Qualitative interviews will be conducted with up to 50% of participants in the ACTIVE group to assess adolescent perspectives of the app and on how the intervention should be disseminated to maximize reach and engagement of high school youth.

CONTROL group participants will be introduced to the NCI webpage and asked to use those resources during the 8-week period and will be scheduled to complete assessments on the same schedule as the ACTIVE group. They will not complete interviews.

Follow-up visits will be conducted 1, 2, 3, and 6 months after the 8 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. high school aged youth (13-19 years old),
2. regular current (past month) e-cig users using nicotine-containing e-cigs at least 1 day/week.
3. want to quit using e-cigarettes.
4. have a smartphone with data/WIFI plan in order to access and utilize the KickNic! app

Exclusion Criteria:

* Those who have non-stable (<2 months) use of anxiolytics, antidepressants, and other psychostimulants or have a history of psychosis or any significant current psychiatric/medical condition that would increase risk will be excluded.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 306 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow Back (self-report) with saliva cotinine (biochemical verification) at 6 month follow up. | 6 month follow up study visit.
  Timeline Follow Back (self-report) determining 7-day point prevalence of e-cigarette use confirmed by saliva cotinine <30ng/mL at 6 month follow up visit.

SECONDARY OUTCOMES:
Timeline Follow Back (self-report) with saliva cotinine (biochemical verification) at End of Treatment (EOT). | EOT (8 weeks).
  Timeline Follow Back (self-report) determining 7-day point prevalence of e-cigarette use confirmed by saliva cotinine <30ng/mL at EOT visit.
Timeline Follow Back (self-report) at EOT, 3, and 6 month follow up | EOT (8 weeks), 3 month follow up, and 6 month follow up.
  Timeline Follow Back (self-report) will be used to determine % days e-cigarette free and continuous abstinence of e-cigarette use at EOT, 3 month, and 6 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, Ph.D., Principal Investigator — Yale University School of Medicine, Dept of Psychiatry
Locations (1):
- Yale University School of Medicine (Connecticut Mental Health Center), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data that underlie results in a publication may be shared with other researchers.